CLINICAL TRIAL: NCT04791605
Title: No Difference in Gait Pattern Between a Cemented and Non-cemented Femur Stem. 45 Prospective Randomized Total Hip Arthroplasty Patients After Acute Cervical Femur Fracture Evaluated After 2 Years
Brief Title: Gait Pattern Between a Cemented and Non-cemented Femur Stem
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cemented and non-cemented stem
Record Dates: First submitted 2021-03-04; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Gait Analysis; Hip Fractures; Hip Arthroplasty; Randomized
MeSH Terms: conditions — Hip Fractures | interventions — Gait Analysis

STUDY DESIGN:
Intervention Model Description: Gait of cemented femur stem of acute cervical collum femoris stem. Gait of non-cemented femur stem of acute cervical collum femoris stem.
Who Masked: Outcomes Assessor
Masking Description: Cemented femur stem Non-cemented femur stem
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gait analysis of cemented total hip (Experimental): Gait analysis of acute collum femoris fracture patient randomized to cemented stem
  Interventions: Other: Gait analysis
- Gait analysis of non-cemented total hip (Experimental): Gait analysis of acute collum femoris fracture patient randomized to non-cemented stem
  Interventions: Other: Gait analysis

INTERVENTIONS:
Other: Gait analysis — Kinematic and kinetic analysis

SUMMARY:
Acute cervical femoral neck fracture patients randomized to either cemented or non-cemented stem. The investigators used gait analysis to evaluate if patients operated with a cemented stem showed more favourable hip kinematics and kinetics when compared with a group of patients operated with a non-cemented stem.

DETAILED DESCRIPTION:
45 patients randomized to receive either a cemented or a non-cemented stem were studied . 2 years after the operation gait analysis was performed with a 16-camera motion capture system together with 2 force-plates. Hip kinematics and kinetics were analysed and 70 subjects served as controls.

ELIGIBILITY:
Inclusion Criteria:

* acute collum femoris fracture

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Gait Analysis with focus on hip kinematics 2 year after total hip arthroplasty | 2 year postop
  Optical tracking system focusing on reflective markers according a model used in gait analysis in order to record degrees of hip angels in 3 planes
Gait Analysis with focus on hip kinetics 2 year after total hip arthroplasty | 2 year postop
  Optical tracking system focusing on reflective markers according a model used in gait analysis together with force plates record hip moments (Nm/kg) in 3 planes

CONTACTS AND LOCATIONS:
Overall Officials: Roland Zügner, Principal Investigator — Göteborg University
Locations (1):
- Roland Zügner, Gothenburg, Sweden

REFERENCES:
- [Derived] Zugner R, Tranberg R, Sharegi B, Karrholm J. Gait pattern in patients treated with a total hip arthroplasty due to an acute displaced cervical neck fracture: a randomised comparison between 29 cases with a cemented femoral stem and 16 cases with an uncemented femoral stem. Hip Int. 2024 May;34(3):421-427. doi: 10.1177/11207000231208099. Epub 2023 Dec 12. PMID 38087800